CLINICAL TRIAL: NCT06864832
Title: Efficacy of Therapeutic Exercise (Mirror Image Exercise) in Adolescent With Chronic Low Back Pain, Through Corrective Postural Changes; Randomized Controlled Trial
Brief Title: Efficacy of Therapeutic Exercise (Mirror Image Exercise) in Adolescent With Chronic Low Back Pain, Through Corrective Postural Changes
Acronym: low back pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Al-Amir Mohamed Hussein, Lecturer of Physical Therapy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BeniSuefU23
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Mirror image exercise is a novel technique that utilizes visual feedback to enhance motor control and body awareness in reducing pain and improving function in individuals with mechanical low back pain.
  Interventions: Other: Mirror image postural exercises
- Control group (Placebo Comparator): Patients in this group received the traditional program of exercises in the form of back muscles stretching exercises and abdominal muscles strengthening exercises.
  Interventions: Other: Back exercises

INTERVENTIONS:
Other: Mirror image postural exercises — Patients will recieve mirror image postural exercise on the 3D postural analysis
  Arms: Study group
Other: Back exercises — Exercises in the form of back muscles stretching exercises and abdominal muscles strengthening exercises.
  Arms: Control group

SUMMARY:
This study will include two groups. The study group will receive mirror-image postural exercise on the 3D postural analysis. The control group will receive a traditional exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Having chronic mechanical low back pain.
* Having a significant translational and/or rotational deformity of the lumbar spine according to the posture index scale.
* Having normal x-ray

Exclusion Criteria:

* Severe cardiovascular disease.
* Previous spinal surgery.
* Abdominal hernia.
* True leg length discrepancy.
* Severe respiratory disease.
* Pregnancy.
* Associated pathologies of lower limbs that may interfere with the posture such as foot, knee, and hip deformities.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 1-3 months
  Measured using Visual analoge scale(VAS)
Postural Alignment | 1-3 months
  Assess through 3D posture assessment
Functional Disability | 1-3 months
  Measured using the Oswestry Disability Index(ODI)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Giza Governorate, Egypt